CLINICAL TRIAL: NCT01780259
Title: A Single-Dose Study to Assess the Pharmacokinetics, Safety, and Tolerability of Intranasally Administered Esketamine in Healthy Subjects
Brief Title: A Study to Assess the Pharmacokinetics, Safety, and Tolerability of Intranasally Administered Esketamine in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100942; ESKETINTRD1001 (Other: Janssen Research & Development, LLC); 2012-004374-25 (EudraCT Number)
Record Dates: First submitted 2013-01-28; First posted 2013-01-31 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
Keywords: Healthy; Esketamine; Pharmacokinetics; Intranasal
MeSH Terms: interventions — Esketamine; Triazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Cohort 1: Treatment A (Experimental): Participants will receive 1 spray of esketamine solution in each nostril once (total dose: 28 mg).
  Interventions: Drug: Esketamine
- Cohort 1: Treatment B (Experimental): Participants will receive 1 spray of esketamine solution in each nostril twice, with 5 minutes interval (total dose: 56 mg).
  Interventions: Drug: Esketamine
- Cohort 1: Treatment C (Experimental): Participants will receive 1 spray of esketamine solution in each nostril thrice, with 5 minutes interval between each repeated sprays (total dose 84 mg).
  Interventions: Drug: Esketamine
- Cohort 1: Treatment D (Experimental): Participants will receive 1 spray of esketamine solution in each nostril thrice, with 10 minutes interval between each repeated sprays (total dose 84 mg).
  Interventions: Drug: Esketamine
- Cohort 2: Treatment D (Experimental): Participants will receive 1 spray of esketamine solution in each nostril thrice, with 10 minutes interval between each repeated sprays (total dose 84 mg).
  Interventions: Drug: Esketamine
- Cohort 3: Treatment E (Experimental): Participants will receive 1 spray of esketamine solution in each nostril, 4 times with 10 minutes interval between each repeated sprays (total dose: 112 mg). Single dose of oral placebo will be administered 5 minutes before the first intranasal spray of esketamine solution.
  Interventions: Drug: Esketamine; Drug: Placebo
- Cohort 3: Treatment F (Experimental): Participants will receive 1 spray of placebo solution in each nostril, 4 times with 10 minutes interval between each repeated sprays (total dose: 112 mg). Single 0.25-mg oral dose of triazolam will be administered 5 minutes before the first intranasal spray of placebo solution.
  Interventions: Drug: Placebo; Drug: Triazolam

INTERVENTIONS:
Drug: Esketamine — 1 spray of 14 percent of esketamine solution (14 mg of esketamine per 100 microlitre) will be administered intranasally by nasal spray pump in each nostril once (Treatment A-total dose: 28 mg), twice with 5 minutes interval (Treatment B-total dose: 56 mg), thrice with 5 minutes interval between each repeated sprays (Treatment C-total dose: 84 mg), thrice with 10 minutes interval between each repeated sprays (Treatment D-total dose: 84 mg) and 4 times with 10 minutes interval between each repeated sprays (Treatment E-total dose: 112 mg). Treatment A, B, C, D will be administered in Cohort 1; Treatment D will be administered in Cohort 2; and Treatment E will be administered in Cohort 3.
  Arms: Cohort 1: Treatment A; Cohort 1: Treatment B; Cohort 1: Treatment C; Cohort 1: Treatment D; Cohort 2: Treatment D; Cohort 3: Treatment E
Drug: Placebo — Single dose of oral placebo will be administered 5 minutes before the first intranasal spray of esketamine solution in the Treatment E of Cohort 3. Placebo solution (solution of water for injection with denatonium benzoate) will be administered intranasally solution by nasal spray pump in the Treatment F of Cohort 3.
  Arms: Cohort 3: Treatment E; Cohort 3: Treatment F
Drug: Triazolam — Single 0.25-mg oral dose of triazolam will be administered 5 minutes before the first intranasal spray of placebo solution in the Treatment F of Cohort 3.
  Arms: Cohort 3: Treatment F

SUMMARY:
The primary purpose of the study is to evaluate the pharmacokinetics (what the body does to the medication) of intranasally (through the nose) administered esketamine in healthy participants.

DETAILED DESCRIPTION:
This is a single-center study with 3 cohorts (groups). Approximately 58 participants will be enrolled in this study. In Cohort 1, approximately 16 participants will be enrolled for up to 78 days and they will receive 4 different single-dose regimens (Treatment A, B, C and D) of intranasal spray of esketamine solution in a crossover manner (participants will be switched from one single-dose regimen to another) and in an open label manner (both the investigator and the participant know the intervention received by the participant). In Cohort 2, approximately 14 participants will be enrolled for up to 35 days and they will receive 1 regimen of intranasal esketamine (Treatment D) in an open label manner. In Cohort 3, approximately 28 participants will be enrolled and they will be randomly assigned to receive either Treatment E (intranasal esketamine spray) or Treatment F (intranasal placebo spray) in a double blind manner (both the investigator and the participant do not know the intervention received by the participant). Safety evaluations will include assessment of adverse events, targeted nasal examinations, laboratory tests, electrocardiogram, physical examination, pulse oximetery, and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Blood pressure between 90 and 145 mmHg systolic and no higher than 90 mmHg diastolic
* A 12-lead electrocardiogram consistent with normal cardiac conduction and function
* Agree to protocol-defined method of contraception
* Comfortable with self-administration of intranasal medication

Exclusion Criteria:

* History of or current clinically significant medical illness including cardiac arrhythmias or other cardiac disease; hematologic disease; coagulation disorders; significant pulmonary disease, including bronchospastic respiratory disease; diabetes mellitus; renal or hepatic insufficiency; thyroid disease; neurologic or psychiatric disease, asthma
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening or at admission to the study center
* Clinically significant abnormal physical examination, vital signs or 12 lead electrocardiogram at screening or at admission to the study center
* Known allergy to heparin or history of heparin-induced thrombocytopenia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2012-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration during a dosing interval (Cmax) of esketamine | Predose, 7 minutes, 12 minutes, 22 minutes, 32 minutes, 40 minutes, 50 minutes, 1 hour, 1.25 hours, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 9 hours, 12 hours, 18 hours, 24 hours
Time to reach the maximum plasma concentration (tmax) of esketamine | Predose, 7 minutes, 12 minutes, 22 minutes, 32 minutes, 40 minutes, 50 minutes, 1 hour, 1.25 hours, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 9 hours, 12 hours, 18 hours, 24 hours
Area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration (AUClast) of esketamine | Predose, 7 minutes, 12 minutes, 22 minutes, 32 minutes, 40 minutes, 50 minutes, 1 hour, 1.25 hours, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 9 hours, 12 hours, 18 hours, 24 hours

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to 78 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium

REFERENCES:
- [Derived] Perez-Ruixo C, Rossenu S, Zannikos P, Nandy P, Singh J, Drevets WC, Perez-Ruixo JJ. Population Pharmacokinetics of Esketamine Nasal Spray and its Metabolite Noresketamine in Healthy Subjects and Patients with Treatment-Resistant Depression. Clin Pharmacokinet. 2021 Apr;60(4):501-516. doi: 10.1007/s40262-020-00953-4. Epub 2020 Oct 31. PMID 33128208